CLINICAL TRIAL: NCT06454331
Title: Effects of Transcranial Direct Cranial Stimulation on Upper Limb Function and Quality of Life in Stroke Patients
Brief Title: tDCS and Upper Extremity Function in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC01900 Tayyab Awan
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: Stroke; upper limb; tDCS
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): The dosage of anodal tDCS will be 20 minutes with an intensity of 2mA. It's administered before exercise therapy sessions over a period of 8 weeks and 3 times a week
  Interventions: Device: Transcranial direct current stimulation
- Sham tDCS Group (Sham Comparator): sham tDCS, task-oriented training (i.e. placing cones on another cone, inserting needles into a box
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — The two key landmarks for EEG electrode placement are the nasion and the inion which are used to define the measurement. Measure the distance between the nasion and the inion along the midline of the head. Divide the nasion-inion distance by two to find the midpoint and mark this midpoint on the scalp along the midline. C3 (left hemisphere of the scalp) and C4 (right hemisphere of the scalp), which are placed 20% of the nasion-inion distance from the midline, and M1, which is placed 10% of this distance from the midline, can be determined using these calculations. From the midpoint marked on the scalp, measure to the left and right sides using the calculated 10% and 20% distances. Mark these points as M1 and its mirror position. Clean the scalp at the marked M1 and its mirror position locations to remove any oils or debris.
  Arms: Active tDCS
Device: Sham transcranial direct current stimulation — it can apply in sitting or supine lying position but it's important to ensure their comfort and safety while facilitating optimal electrode placement and contact with the scalp. Duration of 20 minutes, with Intensity of 0.5mA, and density of 0.02 mA/cm² for 8 weeks on alternative days
  Arms: Sham tDCS Group

SUMMARY:
Research on the effects of Anodal transcranial Direct Current Stimulation (tDCS) on hand dexterity and quality of life in stroke patients is limited. While the highlighted article focuses on Parkinson's disease, it underscores anodal tDCS potential to modulate brain activity and promote neural plasticity, suggesting potential relevance to stroke rehabilitation

DETAILED DESCRIPTION:
tDCS seems like a hopeful way to help stroke patients improve their upper limb function, but there are still some problems and questions that need to be answered. Previous studies have investigated the impact of (tDCS) on upper limb recovery among stroke patients. However, evidence is scarce on the effect of tDCS on hand dexterity and quality of life in stroke patients. Furthermore, these studies have not adequately explored how the severity of stroke influences the efficacy of tDCS on upper limb motor recovery. Additionally, there is a lack of research examining the cumulative effects of tDCS on both upper limb motor recovery and hand dexterity, as well as QoL, particularly concerning stroke severity.

ELIGIBILITY:
Inclusion Criteria:

* Stroke for more than 6 months.
* Age 40-80 years
* Both gender
* National Institutes of Health Stroke Scale (NIHSS) for severity level (Mild (1-4), Moderate (5-15), Moderate to Severe (16-20), Severe (21-42)

Exclusion Criteria:

* Any patient with Upper limb amputation on the effected side, contracture, burn injury that leads to joint limitation and functional limitation.
* Known cases of Multiple Sclerosis and Parkinson and any Musculoskeletal disorder and Cardiopulmonary disorder.
* Any patient with Metallic implants
* Individuals with a history of seizures or epilepsy
* Individuals with Skin allergies on the scalp

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
FMA-Upper Extremity | 8 week
  The Fugl-Meyer Assessment for Upper Extremity (FMA-UE) is a clinical tool for evaluating motor recovery in stroke and neurological conditions affecting the upper limbs and with a sensitivity of 77%, a specificity of 89%. It assesses motor function through tasks like reaching and grasping, scored on a 3-point scale. Higher scores indicate better function, with a maximum score of 66. Clinicians use it to track progress, plan treatment, and assess outcomes in rehabilitation settings
Action Research Arm Test | 8 week
  The Action Research Arm Test (ARAT) is a clinical assessment tool used to evaluate upper limb function and recovery in individuals who have experienced a stroke or other neurological conditions affecting arm movement. The ARAT consists of a series of 19 items/tasks that assess different aspects of upper limb function, including reaching, grasping, gripping, and manipulating objects of various sizes and shapes. The tasks are scored based on the individual's ability to complete them successfully and the quality of movement exhibited during the task. Scores range from 0 to 3. (0=Unable to perform, 1= Partially performs the task, 2= Completes the task with some difficulty and 3= Completes the task without difficulty)

SECONDARY OUTCOMES:
Stroke Specific Quality of Life | 8 week
  The of Stroke Specific Quality of Life (SS-QOL) questionnaire is a tool used to assess the quality of life in individuals who have experienced a stroke. The SS-QOL reveals a sensitivity of 70.0% and a specificity of 75.8%. It measures various domains including physical function, mobility, social participation, emotional well-being, and cognition. The SS-QOL helps clinicians and researchers understand the impact of stroke on a person's overall quality of life and modify interventions accordingly

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, Analytic Code
Time Frame: March 2025 to August 2025